CLINICAL TRIAL: NCT04076189
Title: Time of Initiation of Positive Pressure Ventilation in Non-vigorous Infants Born Through Meconium-stained Amniotic Fluid: a Cross-over Randomized, Control Trial
Brief Title: Time of Positive Pressure Ventilation in Non-vigorous Infants Born Through Meconium-stained Amniotic Fluid
Acronym: MASTIME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Padova (Other)
Collaborators: University of Padova (Other)
Responsible Party: Principal Investigator, Daniele Trevisanuto, Clinical Professor, University Hospital Padova
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UHPadova02/2019
Record Dates: First submitted 2019-08-29; First posted 2019-09-03 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Meconium Aspiration Syndrome; Infant, Newborn, Disease; Neonatal Resuscitation
Keywords: Infant newborn; Meconium Aspiration Syndrome; Neonatal Resuscitation; Positive Pressure Ventilation
MeSH Terms: conditions — Meconium Aspiration Syndrome; Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endotracheal suctioning (Experimental): Procedure includes: Endotracheal intubation-Suctioning-Endotracheal intubation again and initiation of positive pressure ventilation
  Interventions: Procedure: Endotracheal suctioning
- No endotracheal suctioning (Active Comparator): Procedure includes: Initiation of positive pressure ventilation without endotracheal suctioning
  Interventions: Procedure: No endotracheal suctioning

INTERVENTIONS:
Procedure: Endotracheal suctioning — Procedure includes: Endotracheal intubation-Suctioning-Endotracheal intubation again and initiation of positive pressure ventilation
  Arms: Endotracheal suctioning
Procedure: No endotracheal suctioning — Procedure includes: immediate initiation of positive pressure ventilation without intubation and tracheal suctioning
  Arms: No endotracheal suctioning

SUMMARY:
Background: Meconium stained amniotic fluid (MSAF) complicates 3 to 14% of pregnancies, causing meconium aspiration syndrome (MAS) in 5-10% of neonates born. Due to lack of evidence of benefits of endotracheal suctioning at birth in non-vigorous infants, recent neonatal resuscitation guidelines do not recommend it as a routine and they suggest to start ventilation within the first minute of life, which may be critical to reverse asphyxia and stabilize the neonate. There are concerns regarding the safety and efficacy of this change in practice because it is not based on large randomized controlled trials. Besides that, the delay in the beginning of the PPV in these babies has not been previously explored.

Objective: to compare the time of PPV initiation between performing immediate laryngoscopy with intubation and suctioning and performing immediate PPV without intubation in a manikin.

Methods: Level III NICU consultants, residents, and fellows trained in advanced airway management will be randomly assigned to AB arm (endotracheal suction, followed by the procedure without endotracheal suction) and to BA arm (reverse sequence), with a washout period of 6 hour. During each simulation, an external observer will record the time of PPV initiation. The primary outcome measure will be the time of PPV initiation in the endotracheal suction arm compared to the control arm.

DETAILED DESCRIPTION:
Background: Meconium stained amniotic fluid (MSAF) complicates 3 to 14% of pregnancies, causing meconium aspiration syndrome (MAS) in 5-10% of neonates born. Due to lack of evidence of benefits of endotracheal suctioning at birth in non-vigorous infants, recent neonatal resuscitation guidelines do not recommend it as a routine and they suggest to start ventilation within the first minute of life, which may be critical to reverse asphyxia and stabilize the neonate. There are concerns regarding the safety and efficacy of this change in practice because it is not based on large randomized controlled trials. Besides that, the delay in the beginning of the PPV in these babies has not been previously explored.

Objective: to compare the time of PPV initiation between performing immediate laryngoscopy with intubation and suctioning and performing immediate PPV without intubation in a manikin.

Methods: Level III NICU consultants, residents, and fellows trained in advanced airway management will be randomly assigned to AB arm (endotracheal suction, followed by the procedure without endotracheal suction) and to BA arm (reverse sequence), with a washout period of 6 hour. During each simulation, an external observer will record the time of PPV initiation. The primary outcome measure will be the time of PPV initiation in the endotracheal suction arm compared to the control arm.

ELIGIBILITY:
Inclusion Criteria:

* Level III NICU consultants, residents, and fellows trained in advanced airway management will be eligible to participate in the study

Exclusion Criteria:

* No exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2019-09-24 (Actual); Study Completion 2019-09-24 (Actual)

PRIMARY OUTCOMES:
Time of initiation of positive pressure ventilation | 3 minutes

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Azienda Ospedaliera di Padova, University of Padova, Padua
  - University of Padova, Padua

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Wyllie J, Bruinenberg J, Roehr CC, Rudiger M, Trevisanuto D, Urlesberger B. European Resuscitation Council Guidelines for Resuscitation 2015: Section 7. Resuscitation and support of transition of babies at birth. Resuscitation. 2015 Oct;95:249-63. doi: 10.1016/j.resuscitation.2015.07.029. Epub 2015 Oct 15. No abstract available. PMID 26477415
- [Background] Wyckoff MH, Aziz K, Escobedo MB, Kapadia VS, Kattwinkel J, Perlman JM, Simon WM, Weiner GM, Zaichkin JG. Part 13: Neonatal Resuscitation: 2015 American Heart Association Guidelines Update for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2015 Nov 3;132(18 Suppl 2):S543-60. doi: 10.1161/CIR.0000000000000267. No abstract available. PMID 26473001
- [Background] Chettri S, Adhisivam B, Bhat BV. Endotracheal Suction for Nonvigorous Neonates Born through Meconium Stained Amniotic Fluid: A Randomized Controlled Trial. J Pediatr. 2015 May;166(5):1208-1213.e1. doi: 10.1016/j.jpeds.2014.12.076. Epub 2015 Feb 4. PMID 25661412
- [Background] Nangia S, Sunder S, Biswas R, Saili A. Endotracheal suction in term non vigorous meconium stained neonates-A pilot study. Resuscitation. 2016 Aug;105:79-84. doi: 10.1016/j.resuscitation.2016.05.015. Epub 2016 May 30. PMID 27255954
- [Background] Chiruvolu A, Miklis KK, Chen E, Petrey B, Desai S. Delivery Room Management of Meconium-Stained Newborns and Respiratory Support. Pediatrics. 2018 Dec;142(6):e20181485. doi: 10.1542/peds.2018-1485. Epub 2018 Nov 1. PMID 30385640